CLINICAL TRIAL: NCT01492205
Title: A Doctor and Nurse Survey on Using NovoLet® Within the Hospital Practice in Indonesia
Brief Title: NovoLet® Acceptance Study Within the Hospital Practise in Indonesia
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NOPEN3-1887
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Human insulin
  Interventions: Drug: insulin human

INTERVENTIONS:
Drug: insulin human — All subjects were treated with human insulin administered either by using the NovoLet® pre-filled insulin system or the conventional vial and syringe method. Doctors and nurses must personally administer at least 10 insulin doses to each patient under their individual clinical supervision for assessment of the NovoLet® pre-filled insulin system

SUMMARY:
This study is conducted in Asia. The aim of this study is to evaluate the overall acceptance of healthcare professionals (nurses and doctors) to the NovoLet® system used in a hospital environment.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Type 2 diabetes
* Likely to be hospitalised and require insulin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with either type 1 or type 2 diabetes, who were likely to be hospitalised and require insulin therapy in Indonesia
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2005-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Overall acceptance of the NovoLet® system among healthcare professionals (nurses and doctors)

SECONDARY OUTCOMES:
Time taken for the healthcare professionals (nurses and doctors) to teach the patient
Incidence of adverse drug reactions

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Jakarta, Indonesia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com